CLINICAL TRIAL: NCT05915858
Title: Effects of Muscle Energy Technique and Stretching Exercise on Pain, Hip Joint Range of Motion and Function in Working Pregnant Women With Piriformis Syndrome
Brief Title: Muscle Energy Technique and Stretching Exercise in Working Pregnant Women With Piriformis Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0518
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Piriformis Syndrome
Keywords: muscle energy technique,stretching exercise, pain rom
MeSH Terms: conditions — Piriformis Muscle Syndrome | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- muscle energy technique (Experimental): muscle energy technique
  Interventions: Other: muscle energy technique
- stretching exercise (Active Comparator): stretching exercises along with piriformis stretch
  Interventions: Other: stretching exercise

INTERVENTIONS:
Other: muscle energy technique — Group 1: Group 2:
  Muscle energy technique (Reciprocal inhibition) Stretching exercises Static stretching 2 weeks (twelve treatment session) patient supine, the treated leg is placed into flexion at the hip and knee, so that the foot rests on the table lateral to the contra-lateral knee (the leg on the side to be treated is crossed over the other, straight leg).
  * The angle of hip flexion should not exceed 60 degree.
  * The practitioner places one hand on the contra-lateral ASIS to prevent pelvis motion, while the other hand is placed against the lateral flexed knee as this is pushed into resisted abduction to contract piriformis for 7-10 seconds.
  Arms: muscle energy technique
Other: stretching exercise — Following the contraction the practitioner eases the treated side leg into adduction until a sense of resistance is noted; this is held for 10-30 seconds. 2 week (twelve treatment session) practitioner manual stretches the piriformis:
  * The patient lies in supine position the affected leg is placed into flexion at hip and knee so that the foot rests on the table lateral to the contra-lateral knee.
  * The practitioner places one hand over the contra-lateral ASIS to stabilize the pelvis during the exercise and passively abducts and internally rotates the hip medially till the pain is bearable.
  * The process is repeated 3-5 times with a 30
  Arms: stretching exercise

SUMMARY:
Piriformis syndrome is a neuro muscular disorder which occur due to the compression and irritation of the sciatic nerve by the piriformis muscle causing pain, tingling, and numbness in the buttocks and along the sciatic nerve. Muscle energy technique is one of manual technique in which the muscle uses its own energy in the form of isometric contraction to relax the muscle by the autogenic inhibition of reciprocal inhibition. Reciprocal inhibition in muscle energy technique was succeeded in relieving pain and improves flexibility.

DETAILED DESCRIPTION:
Piriformis syndrome is a neuro muscular disorder which occur due to the compression and irritation of the sciatic nerve by the piriformis muscle causing pain, tingling, and numbness in the buttocks and along the sciatic nerve. Muscle energy technique is one of manual technique in which the muscle uses its own energy in the form of isometric contraction to relax the muscle by the autogenic inhibition of reciprocal inhibition. Reciprocal inhibition in muscle energy technique was succeeded in relieving pain and improves flexibility. Stretching exercises improves physical performance ability, prevents injury, reduces muscle pain and increases flexibility. Both muscle energy technique and stretching has shown significant improvement in reducing pain and lower extremity function and increase range of motion.

Randomized clinical trial will be conducted. Sample size of 30 patients will be taken. Non probability convenient sampling will be used.A written consent form will be taken from participants meeting inclusion criteria and will be randomly allocated into two groups, to either the muscle energy technique group or stretching exercises group.Treatment will be given twice a week for twelve treatment session..Numeric pain rating scale will be used to measure the intensity of pain,Lower extremity functional scale will be used to access lower extremity function. Standard goniometer is used to measure hip joint range of motion.All participants in both groups will be evaluated before and after treatment programme.Total duration of study will be six months.Data will be analyzed by using SPSS 25. Key words Muscle energy technique,Stretching exercises,Piriformis syndrome,Pain,Range of motion

ELIGIBILITY:
Inclusion Criteria:

* Age between 25-45 years .
* Tenderness of piriformis muscle.
* Chronic non-specific low back pain patients.
* Women in second trimester of pregnancy
* Multiparous women
* SLR positive below 60 degrees .
* VAS score: 6-10
* Internal rotation of hip less than 45 degrees.

Exclusion Criteria:

* SLR negative test
* Skin allergy
* Pre-eclampsia
* Gestational diabetes mellitus
* Clinical diagnosis of osteoarthritis or history of fracture of lower extremities

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female 25-45age
Enrollment: 30 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-08-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 6months
  Measurement of pain intensity was done by using numeric pain rating scale.it is reliable and valid.subjects were explained about the scale and instructed to indicate the intensity of current,best and worst pain on a scale of zero(no pain) to ten(worst pain)

SECONDARY OUTCOMES:
Measurements of pain Intensity | 6months
  measurement were taking at pre intervention and post intervention after the end of second week intervention.(10) Lower extremity functional scale Lower extremity functional scale is a questionnaire containing twenty question about persons ability to perform everyday task.The LEFS can be used by clinician as a measure of patients initial function,ongoing progress and out come as well as to set functional goals.
  The LEFS has maximum scores of 80 points where lower the score greater disability

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam, MS, Principal Investigator — Riphah International University
Locations (1):
- Lady Willington, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No